CLINICAL TRIAL: NCT04614909
Title: A Phase 0/2 Clinical Trial of Pamiparib in Newly-Diagnosed and Recurrent Glioblastoma Patients
Brief Title: Study of Pamiparib in Newly Diagnosed and rGBM
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nader Sanai (Other)
Collaborators: Barrow Neurological Institute (Other); Ivy Brain Tumor Center (Other); BeiGene (Industry)
Responsible Party: Sponsor-Investigator, Nader Sanai, Deputy Director, Ivy Brain Tumor Center, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-12
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioblastoma Multiforme, Adult
MeSH Terms: conditions — Glioblastoma | interventions — pamiparib; olaparib; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A Newly-diagnosed Glioblastoma Participant treated with Pamiparib (Experimental): Participants undergoing resection for a presumed newly diagnosed glioblastoma (nGBM) will be treated with pamiparib for 4 days prior to surgical resection. Patients who proceed to Phase 2 will receive pamiparib administered orally BID continuously in combination with 6-7 weeks of radiation therapy and pamiparib in combination with TMZ in the maintenance phase.
  Interventions: Drug: Pamiparib; Radiation: Radiation therapy; Drug: Temozolomide
- Arm B Recurrent Glioblastoma Participant treated with Pamiparib (Experimental): Recurrent glioblastoma (rGBM) patients who are scheduled for surgery and expected to receive postoperative fractionated radiotherapy (RT) will be treated with pamiparib for 4 days prior to surgical resection. Patients who proceed to Phase 2 will receive pamiparib administered orally BID continuously in combination with 6-7 weeks of radiation therapy and pamiparib in combination with TMZ in the maintenance phase.
  Interventions: Drug: Pamiparib; Radiation: Radiation therapy; Drug: Temozolomide
- Arm C Recurrent Glioblastoma Participant treated with Olaparib (Experimental): Arm C will be an exploratory arm in recurrent glioblastoma patients (rGBM) treated with Olaparib for 4 days prior to surgical resection. Patients who proceed to Phase 2 will receive olaparib administered orally BID continuously in combination with 6-7 weeks of radiation therapy and pamiparib in combination with TMZ in the maintenance phase.
  Interventions: Drug: Olaparib; Radiation: Radiation therapy; Drug: Temozolomide

INTERVENTIONS:
Drug: Pamiparib — 60mg administered orally BID for 4 days prior to surgical resection
  Arms: Arm A Newly-diagnosed Glioblastoma Participant treated with Pamiparib; Arm B Recurrent Glioblastoma Participant treated with Pamiparib
Drug: Olaparib — 200mg administered orally BID for 4 days prior to surgical resection
  Arms: Arm C Recurrent Glioblastoma Participant treated with Olaparib
Radiation: Radiation therapy — Patients in Phase 2 will receive 6-7 weeks of radiation therapy per standard of care
Drug: Temozolomide — Arm A and Arm B participants after RT is completed, will receive pamiparib in combination with TMZ (newly diagnosed participants). Arm C participants will receive olaparib with TMZ.

SUMMARY:
This is an open-label, single-center Phase 0/2 study that will enroll up to 30 participants with newly diagnosed (N=12) and recurrent glioblastoma (N=18). The trial will be composed of a Phase 0 component (subdivided into Arm A, Arm B, and Arm C), and an Exploratory Phase 2 component. Participants with tumors demonstrating a PK response in the Phase 0 component of the study will graduate to an exploratory Phase 2 component that combines therapeutic dosing of pamiparib plus fractionated radiotherapy (for unmethylated MGMT promoter newly-diagnosed cases), pamiparib plus fractionated radiotherapy (for recurrent cases) or Olaparib plus fractionated radiotherapy (recurrent cases).

ELIGIBILITY:
Inclusion Criteria:

1. Participants undergoing resection for a suspected newly diagnosed glioblastoma who are also planned to follow the standard regimen or;
2. Participants who have had a prior resection of histologically diagnosed glioblastoma (WHO grade IV), defined as participants who have progressed on or following standard therapy, which includes maximal surgical resection, temozolomide, and fractionated radiotherapy. Participants will also need to have radiation planned as part of the post-surgical treatment plan.
3. Participants must have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 2 perpendicular measurements of at least 1 cm.
4. Ability to understand and the willingness to sign a written informed consent document (personally or by the legally authorized representative, if applicable).
5. Participant has voluntarily agreed to participate by giving written informed consent (personally or via legally authorized representative(s), and assent if applicable). Written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.
6. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.
7. Age ≥18 at time of consent
8. Have a performance status (PS) of ≤2 on the Eastern Cooperative Oncology (Group (ECOG) scale (Oken et al. 1982)
9. Ability to swallow oral medications.
10. Participant has adequate bone marrow and organ function
11. Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant who is no longer of childbearing potential due to surgical, chemical, or natural menopause.
12. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to treatment and agreement to use such a method during study participation and for an additional 6 months after the end of treatment administration.
13. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner and for an additional 6 months after the end of treatment administration. Avoid sperm donation for duration of the study and for an additional 6 months after the end of treatment administration.
14. Agreement to adhere to Lifestyle Considerations throughout study duration.
15. Participants who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to Day 1. A washout period of at least 21 days is required between last chemotherapy dose and Day 1 (provided the participant did not receive radiotherapy).
16. Females of child-bearing potential must agree not to breastfeed starting at screening, throughout the study period and for 6 months after final study drug administration

Exclusion Criteria:

1. Current use of coumarin-derived anticoagulant for treatment, prophylaxis or otherwise, that cannot be discontinued prior to surgery. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
2. Pregnancy or lactation.
3. Known allergic reactions to components of the pamiparib capsule/olaparib.
4. Active infection or fever >38.5°C requiring systemic antibiotic, antifungal or antiviral therapy within 4 weeks of Day 1.
5. Known to have active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis.
6. Known active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
7. Any of the following cardiovascular criteria:

   * Current evidence of cardiac ischemia
   * Current symptomatic pulmonary embolism
   * Acute myocardial infarction ≤ 6 months prior to Day 1
   * Heart failure of New York Heart Association Classification III or IV (see Section 13.2) ≤ 6 months prior to Day 1
   * Grade ≥ 2 ventricular arrhythmia ≤ 6 months prior to Day 1
   * Cerebral vascular accident (CVA) or transient ischemic attack (TIA) ≤ 6 months prior to Day 1
8. Participant has myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML
9. Participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
10. Prior therapy with PARP inhibitors.
11. Treatment with another investigational drug or other intervention within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.
12. For Olaparib participants: Use or anticipated need for food and drugs known to be strong or moderate CYP3A inducers or inhibitors ≤10 days (or ≤5 half-lives, whichever is the shorter) prior to day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Systemic plasma PK profile parameters | Day 4 Intra-operative sample
  Total and unbound pamiparib concentration in enhancing and non-enhancing tumor tissue.

SECONDARY OUTCOMES:
Progression-free survival in participants with demonstrated PK effects | 6 months
  6-month progression-free survival (PFS6) rate measured from time of surgery to date of recurrence
Overall survival | 24 months
  Median overall survival
Drug-related toxicity | 24 months
  Incidence of drug-related toxicity
Adverse events | 24 months
  Number of Adverse Events through study completion, assessed up to 24 months
Treatment-emergent adverse events | 24 months
  Number of treatment-emergent adverse events
Deaths | 24 months
  Number and incidence of deaths
Pharmacodynamics (PD) of pamiparib | Day 4 Intra-operative sample
  Quantification of PAR concentration in tumor homogenates

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Director, Ivy Brain Tumor Center
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No